CLINICAL TRIAL: NCT03353506
Title: A Prospective Double Blind Randomized Pilot Study Comparing the Efficacy of Lyophilized Fecal Microbiota Transplantation (FMT) to Lyophilized Sterile Fecal Filtrate in the Management of Recurrent Clostridium Difficile Infection (CDI)
Brief Title: Lyophilized Fecal Transplant vs Lyophilized Fecal Filtrate in Recurrent C Diff Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dina Kao (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor-Investigator, Dina Kao, Medical Doctor, University of Alberta
Organization: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00076309
Record Dates: First submitted 2017-11-06; First posted 2017-11-27 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Enterocolitis; Recurrent Clostridium Difficile Infection
MeSH Terms: conditions — Enterocolitis; Clostridium Infections

STUDY DESIGN:
Intervention Model Description: double blind randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: LFMT and LSFF capsules appear identical. Randomization is performed by lab staff not involved in any aspect of treatment administration or care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LFMT (Active Comparator): Lyophilized fecal microbiota transplant capsules
  Interventions: Biological: LFMT
- LSFF (Experimental): Lyophilized sterile fecal filtrate capsules
  Interventions: Biological: LSFF

INTERVENTIONS:
Biological: LFMT — Lyophilized fecal microbiota transplant
  Arms: LFMT
Biological: LSFF — Lyophilized sterile fecal filtrate
  Arms: LSFF

SUMMARY:
Fecal microbiota transplantation (FMT) for the treatment of recurrent Clostridium difficile infection (RCDI) has traditionally been offered as fecal slurry administered by enema, nasogastric tube or endoscopy. Frozen oral capsules have also shown efficacy. The potential advantage of lyophilized FMT is the relative ease of manufacturing and storage compared with fecal slurry.

Sterile fecal filtrate has previously been shown to prevent Clostridium difficile infection (CDI) recurrence, suggesting that live bacteria may not be needed. This study will compare lyophilized sterile fecal filtrate (LSFF) with lyophilized FMT (LFMT) in the treatment of recurrent Clostridium difficile infection (RCDI).

DETAILED DESCRIPTION:
This prospective double blind randomized pilot study will enroll 40 subjects with recurrent Clostridium difficile infection in a 1:1 ratio to receive either LSFF or LFMT by capsules.

Subjects will receive 15 capsules at week 0 and be assessed at Weeks 1, 4, 12 and 24. If treatment fails, subjects will be given open label LFMT from the same donor. If treatment fails again, another FMT will be offered and the form and route of FMT delivery will be at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. at least 3 episodes of recurrent CDI, with each episode defined as 3 or more unformed stools in 24 hours associated with positive Clostridium difficile toxin, each occurring within 3 months of each other.
2. CDI under symptomatic control with 3 or fewer unformed stools in 24 hours for at least 2 consecutive days prior to treatment
3. Ability to provide informed consent.
4. Females and males must agree to use effective contraception for the duration of the study as applicable

Exclusion Criteria:

1. Complicated CDI defined as WBC >35, significant abdominal pain and distention, evidence of toxin megacolon or pseudomembraneous colitis, hypotension defined as systolic blood pressure <90 mmHg unresponsive to fluid resuscitation, end organ failure, or requiring admission to intensive care.
2. Chronic diarrheal illness such as irritable bowel syndrome or inflammatory bowel disease unless under control or in remission of 3 months prior to enrollment.
3. Taking or planning to take an investigational drug within 3 months of enrollment.
4. Immunosuppression
5. Chemotherapy or radiation therapy
6. oropharyngeal or significant esophageal dysphagia
7. Ileus or small bowel obstruction
8. Subtotal colectomy
9. Pregnancy or planning to become pregnant within 3 months of enrollment
10. Breastfeeding or planning to breastfeed during the trial
11. Active infection requiring antibiotic therapy.
12. Life expectancy <6 months -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Resolution of RCDI | 8 weeks
  Proportion of subjects without RCDI

SECONDARY OUTCOMES:
Resolution of RCDI | 24 weeks
  Proportion of subjects with sustained cure
Serious Adverse Events | 8 weeks
  Mortality directly attributable to CDI or treatment
Serious Adverse Events | 8 weeks
  Infection directly attributable to treatment
Minor Adverse Events | 1 week
  nausea
Minor Adverse Events | 1 week
  vomiting
Minor Adverse Events | 1 week
  abdominal pain
Difficulty in swallowing capsules | 1 week
  Reported by subjects as ranging between none, moderate or severe

CONTACTS AND LOCATIONS:
Overall Officials: Dina Kao, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No